CLINICAL TRIAL: NCT03992885
Title: Combination Therapy With Ectiecinib, Pemetrexed and Platinum in Patients With Metastatic Non-squamous Non-small Cell Lung Cancer With EGFR Mutations Who Did Not Progress After Pemetrexed in Combination With Platinum-based Chemotherapy:a Single-arm, Open, Multicenter Clinical Study.
Brief Title: Clinical Study of Combination Therapy With Ectiecinib, Pemetrexed and Platinum in Patients With Metastatic Non-squamous Non-small Cell Lung Cancer With EGFR Mutations.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2019161
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: the combination therapy of targeted therapy and chemotherapy; metastatic non-squamous non-small cell lung cancer with EGFR mutations; ectiecinib
MeSH Terms: interventions — icotinib; Pemetrexed; Platinum

STUDY DESIGN:
Intervention Model Description: EGFR-positive patients with metastatic non-squamous non-small cell lung cancer who did not progress after pemetrexed combined with platinum chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy with ectiecinib, pemetrexed and platinum (Experimental): ectinib 125mg/ tablet, one tablet at a time, three times a day, take orally;Pemetrexed 500mg/m2, intravenous infusion, day 1;Carboplatin AUC6/ Cisplatin 75mg/m2,intravenous infusion, day 1,21 days for a cycle, a total of 6 cycles.Maintenance therapy: ectinib: ectinib 125mg/ tablet, one tablet at a time, three times a day, take orally, pemetrexed 500mg/m2,d intravenous infusion, day 1,21 days for a cycle
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Intervention: Drug: Icotinib Ectinib 125mg/ tablet, one tablet at a time, three times a day, take orally
  Intervention: Drug: Carboplatin/ Cisplatin Pemetrexed 500mg/m2, intravenous infusion, day 1;Carboplatin AUC6/ Cisplatin 75mg/m2,intravenous infusion, day 1,21 days for a cycle
  Other Names: Pemetrexed; platinum

SUMMARY:
This single-arm, open, multicenter clinical study is going to evaluate the efficacy and safety of combination therapy with ectiecinib, pemetrexed and platinum in patients with metastatic non-squamous non-small cell lung cancer with EGFR mutations who did not progress after pemetrexed in combination with platinum-based chemotherapy.

DETAILED DESCRIPTION:
The positive rate of EGFR mutations in lung adenocarcinoma patients is about 50% in both Asian population and China.Domestic and international clinical studies have found that targeted therapy combination chemotherapy can prolong the overall survival of patients with EGFR mutations, and a large number of class 2A evidences have been recommended.The 2018 CSCO lung cancer guidelines recommend EGFR-TKIs combined with chemotherapy for first-line treatment of advanced EGFR mutant NSCLC (grade II recommended).The independently developed ectinib in China, belong to EGFR-TKIs as gefitinib and erlotinib . The results of phase III clinical trial (ICOGEN) showed that the efficacy of ectinib and gefitinib was similar, but in terms of safety, the adverse reactions of the ectinib group were significantly lower than that of the gefitinib group, and the difference between the two groups was statistically significant.Targeted combination chemotherapy has relatively large side effects, which will increase chemotherapy-related side effects, mainly hematological toxicity. Foreign studies suggest that combination therapy may be more suitable for patients with good basic state.Based on previous studies, this study is going to use the strategy of short-term induction chemotherapy and drug sensitivity platform to find the most suitable patients for combined therapy.

This single-arm, open, multicenter clinical study is going to evaluate the efficacy and safety of combination therapy with ectiecinib, pemetrexed and platinum in patients with metastatic non-squamous non-small cell lung cancer with EGFR mutations who did not progress after pemetrexed in combination with platinum-based chemotherapy.

Patients received two cycles of chemotherapy with pemetrexed/platinum before enrolling, followed by ectinib: ectinib 125mg/ tablet, one tablet at a time, three times a day, take orally, until disease progression;Pemetrexed 500mg/m2, intravenously administered on day 1;Carboplatin AUC6/ Cisplatin 75mg/m2,intravenously on day 1,21 days for a cycle, a total of 6 cycles.Maintenance therapy: ectinib: ectinib 125mg/ tablet, one tablet at a time, three times a day, take orally, pemetrexed 500mg/m2, intravenously on day 1,21 days for a cycle, until disease progression.Make detailed records of toxic and side effects during medication.The efficacy was evaluated using RESIST standard after every 2 cycles of the treatment, the regimen will continue until the disease progression or the appearance of not tolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75;
2. Expected survival is at least 12 weeks;
3. Metastatic non-squamous non-small cell lung cancer with EGFR mutations confirmed by histological or cytological examination;
4. Received two cycles of pemetrexed/platinum chemotherapy with no progress (efficacy was evaluated as SD or PR);
5. Tumor specimens must be provided before patients receive ectinib combined chemotherapy to complete the EGFR gene test. There is no need to clarify the EGFR mutation status before the initial pemetrexed/platinum chemotherapy;
6. Volunteers who participate in exploratory studies need provide tumor samples for the laboratory to complete the study on anti-tumor drug sensitivity of microfluidic chip technology;
7. Volunteers who participate in exploratory studies need provide blood samples to complete the analysis of blood biomarkers and disease progression/anti-tumor efficacy, tolerance and safety of drugs;
8. 0-1 ECOG score;
9. Patients may have a history of brain parenchymal metastasis, and local treatment (surgery and/or radiotherapy) is required for good control of symptoms, and hormone maintenance therapy is not required;
10. According to RECIST criteria 1.1, there is at least one measurable lesion that has not been irradiated:1) if there is at least one measurable lesion, and if there is only one lesion, the nature of new organisms at the lesion site must be confirmed by cytology or histology;2) for patients with at least one lesion diameter that can be accurately measured by any of the following methods, computed tomography (CT) or magnetic resonance (MRI) of chest or abdomen, the diameter of which should be at least 20mm by conventional methods or at least 10mm by spiral CT;
11. The level of organ function must meet the following requirements:1) bone marrow: median granulocyte absolute count (ANC) ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥9 g/dL;2) liver: serum bilirubin ≤1.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5 times the upper limit of normal value (ALT ≤ 5 times the upper limit of normal value if there is liver metastasis);3) upper limit of serum creatinine <1.5 times normal value;Creatinine clearance ≥50 mL/min (calculated by cockroft-gault10 formula) for patients with low body weight or patients with significantly different values calculated by the two formulas, it is recommended to measure creatinine clearance by other methods, such as EDTA method, inulin clearance method, or 24-hour urinalysis.4) international standardized ratio of prothrombin time (INR) ≤1.5 and partial thrombin time (APTT) ≤1.5 upper limit of normal value in patients who have not received anticoagulation therapy.Patients receiving full or parenteral anticoagulant therapy can enter the clinical trial as long as the dose of anticoagulant is stable for at least 2 weeks before entering the clinical study and the results of coagulation test are within the limits of local treatment.
12. Women of reproductive age must have negative serum pregnancy test results within 7 days prior to treatment;All enrolled patients (male or female) should take adequate barrier contraception during and within 4 weeks after treatment;
13. Patients must be able to understand and sign informed consent voluntarily, prior to any trial procedures.

Exclusion Criteria:

1. Previous EGFR-TKIs targeted drug therapy;
2. Allergic history or hypersensitivity history of patients to active ingredients or non-active excipients of experimental drugs, drugs with chemical structure similar to experimental drugs, or similar drugs of experimental drugs;
3. Known CYP inhibitors or inducers, such as phenytoin, carbamazepine, rifampicin, barbiturate, or st. John's wort, are currently being used (or cannot be discontinued within 1 week prior to the first administration);
4. Patient's organs and systems:1) patients with brain/meningeal metastasis (except those who do not need hormone maintenance therapy after local treatment for brain parenchymal metastasis is controlled);2) having had interstitial lung disease, drug-induced interstitial disease, radiation pneumonia requiring hormone therapy, or any active interstitial lung disease with clinical evidence, and having had idiopathic pulmonary fibrosis on CT scan at baseline;Uncontrolled massive pleural or pericardial effusion;3) evidence of serious or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, heart, liver or kidney disease), as determined by the investigator;4) any unstable systemic disease (including active >CTCAE grade 2 clinical severe infection, grade 4 hypertension, unstable angina pectoris, congestive heart failure, human immunodeficiency virus (HIV) infection, liver, kidney or metabolic disease);5) any other malignancy (other than fully cured cervical carcinoma in situ or basal or squamous cell skin cancer) within 5 years;6) a clear history of neurological or psychiatric disorders, including epilepsy or dementia;7) patients with a history of allogeneic organ transplantation;Patients who underwent major surgery or suffered severe trauma within 4 weeks prior to first administration;8) more than 30% of the experimental drugs received extensive radiotherapy or bone marrow radiotherapy within 4 weeks before the first administration;
5. Any conditions that affect the swallowing or absorption of medications, such as refractory nausea and vomiting, inability to swallow test medications, history of any type of gastrointestinal tract resection or surgery;
6. Pregnant or lactating females (males and females participating in this study must take adequate barrier contraceptive measures during and within 4 weeks after the end of the study);
7. Existing substance abuse and medical, psychological or social conditions that may interfere with patients participating in or evaluating research results;
8. Any unstable or potentially compromising patient safety and compliance with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 5 years
  PFS was defined as the length of time from the date of randomization to the date of disease progression was first observed (as determined by imaging), and the number of days from the date of randomization to death if the patient died of other causes before the disease progression.
Overall survival | 5 years
  OS was defined as the length of time from the date of randomization to death from any cause.Patients who are alive as of the date of analysis will have their last contact as the cut-off date.

SECONDARY OUTCOMES:
Objective response rate | 5 years
  Objective response rate was defined as the percentage of patients whose tumor shrinkage has reached a certain point and remains there for a certain period of time, including cases of complete response and partial response.
Adverse Events | 5 years
  Adverse events are unforeseeable medical conditions or deterioration of pre-existing medical conditions that occur during or after the use of a drug, regardless of whether it is related to the drug in question.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Chen, M.D., Principal Investigator — Department of Pulmonary Medical Oncology, Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Pulmonary Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Result] Mehic B, Duranovic Rayan L, Bilalovic N, Dohranovic Tafro D, Pilav I. Lung adenocarcinoma mimicking pulmonary fibrosis-a case report. BMC Cancer. 2016 Sep 13;16(1):729. doi: 10.1186/s12885-016-2763-6. PMID 27619516
- [Result] Inoue A, Kobayashi K, Maemondo M, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Updated overall survival results from a randomized phase III trial comparing gefitinib with carboplatin-paclitaxel for chemo-naive non-small cell lung cancer with sensitive EGFR gene mutations (NEJ002). Ann Oncol. 2013 Jan;24(1):54-9. doi: 10.1093/annonc/mds214. Epub 2012 Sep 11. PMID 22967997